CLINICAL TRIAL: NCT05725161
Title: Acceptance and Commitment Therapy Supplemented With Psychoeducation for Improving Mental Health of Depressed Individuals Living With Spinal Cord Injury Sustained Within 5 Years
Brief Title: Acceptance and Commitment Therapy for Depressed Individuals Living With Spinal Cord Injury Sustained Within 5 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Paralyzed Veterans of America (Other)
Responsible Party: Principal Investigator, Areum Han, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3191
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Depression; Spinal Cord Injuries
Keywords: Acceptance and Commitment Therapy; Anxiety; Depression; Grief; Mindfulness; Resilience; Self-compassion; Stress; Spinal cord injuries; Quality of life
MeSH Terms: conditions — Depression; Spinal Cord Injuries; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment therapy (ACT) group (Experimental): 8 weekly ACT sessions individually guided by a trained coach through Zoom videoconferencing with psychoeducation materials provided
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Wait-list control group with psychoeducation materials provided (Other): Care as usual with psychoeducation materials provided during the study period and ACT sessions provided after the study period ends
  Interventions: Behavioral: Wait-list control group with psychoeducation materials provided

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy (ACT) — Participants assigned to the ACT group will receive 8 weekly individual ACT sessions guided by a coach for one hour per week over 8 weeks through Zoom videoconferencing with psychoeducation materials provided.
  Arms: Acceptance and commitment therapy (ACT) group
Behavioral: Wait-list control group with psychoeducation materials provided — The wait-list control group will receive care as usual with psychoeducation materials provided during the study period and receive ACT sessions after the study period ends
  Arms: Wait-list control group with psychoeducation materials provided

SUMMARY:
This randomized controlled trial aims to assess effects of videoconferencing acceptance and commitment therapy (ACT) on mental health outcomes in individuals living with spinal cord injuries (SCI). A total of 34 individuals living with SCI sustained within 5 years and experiencing depressive symptoms will be recruited and randomly assigned to either the ACT group or the wait-list control group. The ACT group will receive 8 weekly individual ACT sessions guided by a coach through videoconferencing. The wait-list group will receive ACT sessions after the study period ends. We will provide psychoeducation materials related to SCI as supplemental resources to both groups. Mental health outcomes using self-reported questionnaires will be collected at pretest, posttest, and 2-month follow-up. Exploratory hypotheses are that the group undergoing the ACT intervention supplemented with psychoeducation will show improvements in mental health outcomes (e.g., depression) and ACT processes (e.g., psychological flexibility) at posttest and 2-month follow-up, compared to the wait-list control group provided with psychoeducation materials alone. Interviews will be conducted at posttest to explore the participants' experiences in ACT.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess effects of videoconferencing acceptance and commitment therapy (ACT) on mental health outcomes in individuals living with spinal cord injuries (SCI). A total of 34 individuals living with SCI sustained within 5 years and experiencing depressive symptoms will be recruited and randomly assigned to either the ACT group or the wait-list control group. The ACT group will receive 8 weekly individual ACT sessions guided by a coach through videoconferencing. The wait-list group will receive ACT sessions after the study period ends. We will provide psychoeducation materials related to SCI as supplemental resources to both groups. Mental health outcomes using self-reported questionnaires will be collected at pretest, posttest, and 2-month follow-up. Exploratory hypotheses are that the group undergoing the ACT intervention supplemented with psychoeducation will show improvements in depression (primary outcome), secondary mental health outcomes (e.g., anxiety, stress, and grief), and ACT processes (e.g., psychological flexibility) at posttest and 2-month follow-up, compared to the wait-list control group provided with psychoeducation materials alone. Interviews will be conducted at posttest to explore the participants' experiences in ACT.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults (aged 18 years or older) living with spinal cord injuries sustained within 5 years
* having at least mild depression measured by the Patient Health Questionnaire-9
* having a computer or a smartphone and internet access at home

Exclusion Criteria:

* having cognitive deficits or language barriers that might impede study participation
* having suicidal attempts within 6 months;
* having a prior experience with acceptance and commitment therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline to immediately after the intervention and 2 month follow-up on the Patient Health Questionnaire-9 | Change from baseline to immediately after the intervention and 2 month follow-up
  The Patient Health Questionnaire-9 is a 9-item questionnaire assessing depressive symptoms on a scale of 0 to 3. Scores range from 0 to 27. Higher scores indicate greater symptomatology in depression.

SECONDARY OUTCOMES:
Change from baseline to immediately after the intervention and 2 month follow-up on the Generalized Anxiety Disorder-7 | Change from baseline to immediately after the intervention and 2 month follow-up
  The Generalized Anxiety Disorder-7 is a 7-item questionnaire assessing anxiety on a scale of 0 to 3. Scores range from 0 to 21. Higher scores indicate greater anxiety.
Change from baseline to immediately after the intervention and 2 month follow-up on the Perceived Stress Scale | Change from baseline to immediately after the intervention and 2 month follow-up
  The Perceived Stress Scale is a 10-item questionnaire assessing stress on a scale of 0 to 4. Scores range from 0 to 40. Higher scores indicate greater stress.
Change from baseline to immediately after the intervention and 2 month follow-up on the World Health Organization Quality of Life - Psychological health component | Change from baseline to immediately after the intervention and 2 month follow-up
  World Health Organization Quality of Life - Psychological health component has 6 items measuring psychological quality of life on scale of 1 to 5. Scores range from 6 to 30. Higher scores denote higher quality of life in terms of psychological health.
Change from baseline to immediately after the intervention and 2 month follow-up on the Spinal Cord Injury-Quality of Life (SCI-QOL) Grief and Loss Short form | Change from baseline to immediately after the intervention and 2 month follow-up
  SCI-QOL Grief and Loss Short form has nine items assessing grief and loss due to SCI on a scale of 1 to 5. Scores range from 9 to 45, and higher scores indicate more grief and loss.
Change from baseline to immediately after the intervention and 2 month follow-up on the SCI-QOL Resilience Short form | Change from baseline to immediately after the intervention and 2 month follow-up
  SCI-QOL Resilience Short form has eight items assessing resilience on a scale of 1 to 5. Scores range from 8 to 40, and higher scores indicate greater resilience.
Change from baseline to immediately after the intervention and 2 month follow-up on the Self-Compassion Scale- Short Form | Change from baseline to immediately after the intervention and 2 month follow-up
  Self-Compassion Scale- Short Form is a 12-item self-report questionnaire assessing self-compassion on a scale of 1 to 5. Scores range from 12 to 60. Higher scores indicate higher levels of self-compassion.
Change from baseline to immediately after the intervention and 2 month follow-up on the Action and Acceptance Questionnaire-II | Change from baseline to immediately after the intervention and 2 month follow-up
  Action and Acceptance Questionnaire -II is a 7-item self-report questionnaire measuring psychological flexibility on a scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate poor psychological flexibility.
Change from baseline to immediately after the intervention and 2 month follow-up on the Cognitive Fusion Questionnaire | Change from baseline to immediately after the intervention and 2 month follow-up
  Cognitive Fusion Questionnaire -7 is a 7-item self-report questionnaire measuring cognitive fusion on scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate greater levels of cognitive fusion.
Change from baseline to immediately after the intervention and 2-month follow-up on the Engaged Living Scale | Change from baseline to immediately after the intervention and 2 month follow-up
  Engaged Living Scale -9 is a 9-item self-assessment instrument that measures clarity and engagement with personal values and life fulfillment on a scale of 1 to 5. The total scores range from 9 to 45, and higher scores indicate increased clarity and engagement with personal values and greater life fulfillment.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han A, Wilroy JD, Yuen HK, Jenkins J, Hawkins J. Videoconference-delivered acceptance and commitment therapy for depressed individuals with spinal cord injury sustained within the past 5 years: A pilot randomized controlled trial. Rehabil Psychol. 2025 Dec 1. doi: 10.1037/rep0000642. Online ahead of print. PMID 41325142